CLINICAL TRIAL: NCT03018899
Title: Comparison of Paravertebral Block Versus Epidural Anesthesia for Surgical Anesthesia of Percutaneous Nephrolithotomy
Brief Title: Paravertebral Block Versus Epidural Anesthesia for Percutaneous Nephrolithotomy
Acronym: PVB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Vice Director, Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PVB-TJ
Record Dates: First submitted 2016-10-13; First posted 2017-01-12 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Kidney Calculi
Keywords: paravertebral block; ultrasound; percutaneous nephrolithotomy; postoperative pain
MeSH Terms: conditions — Kidney Calculi; Pain, Postoperative | interventions — Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- paravertebral block (Experimental): patients received ultrasound guided two-segment paravertebral block for percutaneous nephrolithotomy
  Interventions: Procedure: paravertebral block
- Epidural (Active Comparator): patients received thoracic epidural anesthesia for percutaneous nephrolithotomy
  Interventions: Procedure: epidural anesthesia

INTERVENTIONS:
Procedure: paravertebral block — Ultrasound guided two-segment paravertebral block
  Arms: paravertebral block
Procedure: epidural anesthesia — thoracic epidural anesthesia
  Arms: Epidural

SUMMARY:
This prospective, randomized study is aimed to assess the efficacy and safety of paravertebral block compared to epidural anesthesia for percutaneous nephrolithotomy. The investigators suppose that paravertebral block is not inferior in controlling the perioperative pain for percutaneous nephrolithotomy compared to epidural block.

DETAILED DESCRIPTION:
Background: Percutaneous nephrolithotomy (PCNL) is generally performed under general or neuraxial anesthesia. The investigators have reported three patients who were at high risk of both general anesthesia and neuraxial anesthesia received percutaneous nephrolithotomy with ultrasound guided paravertebral block. Then，The investigators performed ultrasound guided paravertebral block for 45 patients who received percutaneous nephrolithotomy successfully. The investigators' impression is that paravertebral block is as effective as epidural anesthesia for surgical anesthesia of percutaneous nephrolithotomy.

Objectives:To assess the efficacy and safety of paravertebral block compared to epidural anesthesia for surgical anesthesia of percutaneous nephrolithotomy.

Methods: Fifty adult patients undergoing elective percutaneous nephrolithotomy will be randomized to receive ultrasound guided paravertebral block or epidural anesthesia. The primary outcome will be the pain score 12h postoperation. The secondary outcomes will include: time spent to perform block, dose of intraoperative opioids, rate of hypotension need for vasoconstrictors, muscle Power Grading of the lower legs at the end of the operation, anus exhaust time, opioid consumption postoperation, postoperative PONV score and the frequency of vomiting , hospitalization duration and patient satisfaction.

Clinical Implications: Ultrasound guided paravertebral block could be an equally effective and safe alternative to epidural block for surgical anesthesia of percutaneous nephrolithotomy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo first stage percutaneous nephrolithotomy
* Informed consent

Exclusion Criteria:

* BMI>35
* Coagulopathy, on anticoagulants
* History of surgery on spine
* Spine deformity
* A known allergy to the drugs being used
* Tumor or infection at the site of puncture
* inability to provide adequate informed consent
* refusal to participate in the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
pain score 12h post operation | 12 hours postoperation

SECONDARY OUTCOMES:
time spent to perform block | during block
dose of intraoperative opioids | during operation
rate of hypotension | during operation
Muscle Power Grading of the lower legs at the end of the operation | 12 hours postoperation
opioid consumption postoperation | 12 hours postoperation
postoperative PONV score and the frequency of vomiting | 24 hours postoperation
Hospitalization duration | 10 days postoperation
Patient satisfaction | one day before discharge
  Patient satisfaction will be evaluated by 5-point Likert scal

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, Doctor, Study Director — Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
For patient's privacy